CLINICAL TRIAL: NCT06332482
Title: Complete Digital Workflow for Construction of Full Arch Implant Supported Screw Retained Restoration :occlusal Accuracy of Different Techniques Used to Record Maxillo-mandibular Relationship(Crossover Study)
Brief Title: Complete Digital Workflow for Construction of Full Arch Implant Supported Screw Retained Restoration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: M0303023RP
Record Dates: First submitted 2023-10-10; First posted 2024-03-27 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: digital impressions will be made for each patient,3 technique will be used to determine intermaxillary relation. Occlusal prematurties of final prosthesis will compared using occlusense device and all patients will be followed up for one year
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Active Comparator): Patients who will use surgical stent in recording the digital Jaw relation
  Interventions: Device: Implant supported screw retained prosthesis
- Group 2 (Active Comparator): Patients who will use acrylic complete denture in recording the digital Jaw relation
  Interventions: Device: Implant supported screw retained prosthesis
- Group 3 (Active Comparator): Patients who will use mandibular stent in recording the digital Jaw relation
  Interventions: Device: Implant supported screw retained prosthesis

INTERVENTIONS:
Device: Implant supported screw retained prosthesis — All patients will receive six maxillary and mandibular implants for full arch screw retained prosthesis

SUMMARY:
This study will compare the occlusal accuracy of different techniques for recording maxillomandibular relationships in a Complete digital workflow to construct full arch implant-supported screw-retained restoration.

ELIGIBILITY:
Inclusion Criteria:

* • Inclusion criteria: i- complete maxillary and mandibular edentulous arches ii- residual alveolar ridges covered with healthy firmly attached mucosa. iii- Angel's class I maxillo-mandibular relationship and iv- Adequate bone height and width for placement of standard diameter implants.

Exclusion Criteria:

* History of drug administration that interfere with bone quality ii- Surgical contraindication (patients under anticoagulant ,immunosuppressive drugs, chemotherapy and irradiation therapy) iv- tempromandibular or myoneurological disorders.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
measurement of occlusal prematurity | one year
  Occlusal prematureties of final prosthesis will be measured using occlusense device
prosthestic complications | one year
  prosthetic complications will be recorded for all patients and statistically analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University ,Faculty of dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No